CLINICAL TRIAL: NCT04939909
Title: Botulinum Toxin Relieves Anxiety, Depression and Sleep Disorderes in Patients With Blepharospasm
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-487
Record Dates: First submitted 2021-06-01; First posted 2021-06-25 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2021-07

CONDITIONS: Blepharospasm
MeSH Terms: conditions — Blepharospasm | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients treated with Botulinum toxin type A (Other): Patients were treated with Botulinum toxin type A
  Interventions: Drug: Botulinum toxin type A

INTERVENTIONS:
Drug: Botulinum toxin type A — Patients were treated with Botulinum toxin type A applications on the Orbicularis oculi and glabellar complex

SUMMARY:
Blepharospasm (BSP) is a chronic, idiopathic, recurrent and progressive disease, which mostly occurs in both eyes. It is mainly manifested as involuntary spasm of muscles around the eyes, leading to uncontrollable narrowing or even closure of blepharospasm. Although there is no pain in BSP patients, it can cause social or psychological dysfunction, make patients feel difficult in driving, reading and working, and seriously affect the social, work and life of patients.

Depression and anxiety are common and harmful mental disorders. At present, less than 40% of patients with depression can get effective treatment. Using simple and effective screening tools can effectively improve the detection rate of depression, so that patients can get timely and effective treatment. It is also an effective measure to prevent suicide.

Botulinum toxin type A (BTX-A) has achieved gratifying results in the treatment of dyskinesia. It has been confirmed that BTX-A has a significant effect on BSP. The effective rate is 70% - 90%. About 50% of the patients can regain normal or near normal visual function. At present, no prospective studies have explored this association between blepharospasm and depression / anxiety, and whether BTX-A can improve this mood disorder. Therefore, our research goal is to further study the relationship between blepharospasm and depression / anxiety, sleep in a prospective way, and to determine whether BTX-A treatment will affect depression / anxiety symptoms, so as to provide more theoretical basis for clinical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with blepharospasm who received botulinum toxin injection therapy
* All patients must have had the symptoms of blepharospasm for over six months

Exclusion Criteria:

* Glaucoma
* Age-related macular degeneration
* Visual acuity of 20/200 or worse
* Chronic obstructive pulmonary disease
* Cardio cerebral diseases, psychosis
* Loss of limb
* Connective tissue diseases
* Dialysis dependence
* Anyone who was unable to cooperate with the examinations

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-07-12 (Actual); Primary Completion 2021-12-24 (Actual); Study Completion 2022-07-15 (Estimated)

PRIMARY OUTCOMES:
Change from baseline blepharospasm evaluation at 3 months | Through study completion, 3 months.
  Patients will evaluated the Jankovic Rating scale (JRS)，the total score of JRS is 8, and a change of 2 points in the JRS is clinically meaningful.

SECONDARY OUTCOMES:
Change from baseline depression evaluation at 3 months | Through study completion, 3 months.
  Patients will evaluated the personal Health Questionnaire Depression Scale (PHQ-8) with a total score of 24, cut-points of 5, 10, and 15 represent mild, moderate, and severe levels of depressive symptoms.
Change from baseline anxiety evaluation at 3 months | Through study completion, 3 months.
  Patients will evaluated the Generalized Anxiety Disorder 7-item scale (GAD-7) questionnaires with a total score of 21, cut-points of 5, 10, and 15 represent mild, moderate, and severe levels of anxiety symptoms.

OTHER OUTCOMES:
Change from baseline sleep disorders evaluation at 3 months | Through study completion, 3 months.
  Patients will evaluated the Athens insomnia scale (AIS) questionnaires, the severity criteria of the AIS are capable of categorizing insomnia severity as follows: absence of insomnia (0-5), mild insomnia (6-9), moderate insomnia (10-15), and severe insomnia (16-24).

CONTACTS AND LOCATIONS:
Overall Officials: Juan Ye, Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University; Huina Zhang, Study Director — Second Affiliated Hospital, School of Medicine, Zhejiang University; Qi Gao, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University; Jiajun Xie, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Juan Ye, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided